CLINICAL TRIAL: NCT00006027
Title: A Phase III Study of Adjuvant Postoperative Irradiation With or Without Cisplatin/Taxol Chemotherapy Following TAH/BSO for Patients With Endometrial Cancer
Brief Title: Comparison of Radiation Therapy With or Without Combination Chemotherapy Following Surgery in Treating Patients With Stage I or Stage II Endometrial Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: RTOG-9905; CDR0000068040; GOG-0194
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2013-08

CONDITIONS: Endometrial Cancer
Keywords: stage I endometrial carcinoma; stage II endometrial carcinoma; endometrial adenocarcinoma; endometrial adenosquamous cell carcinoma; endometrial adenoacanthoma; endometrial clear cell carcinoma; endometrial papillary serous carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Cisplatin; Paclitaxel; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin
Drug: paclitaxel
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor tissue. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if radiation therapy is more effective with or without combination chemotherapy for endometrial cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with or without combination chemotherapy following surgery in treating patients who have stage I or stage II endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the relapse-free survival in patients with stage I or II endometrial cancer treated with adjuvant radiotherapy with or without cisplatin and paclitaxel after total abdominal hysterectomy and bilateral salpingo-oophorectomy.
* Compare the patterns of recurrence and the acute and late toxicity profiles associated with these treatment regimens in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease stage (IC-IIA vs IIB). Patients are randomized to one of two treatment arms.

* Arm I: Within 8 weeks after surgery, patients receive radiotherapy once daily 5 days a week for 5.5 weeks.
* Arm II: Within 8 weeks after surgery, patients receive radiotherapy as in arm I concurrently with cisplatin IV over 2-4 hours on days 1 and 28. After completion of radiotherapy, patients receive paclitaxel IV over 3 hours followed by cisplatin IV over 2-4 hours on days 56, 84, 112, and 140.

Patients are followed every 3 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 436 patients (218 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed uterine confined endometrioid endometrial adenocarcinoma with one of the following:

  * Grade 2 or 3 carcinoma with more than 50% myometrial invasion (stage IC and IIA)
  * Grade 2 or 3 carcinoma with stromal invasion of the cervix (stage IIB)
* No grade I adenocarcinoma
* Less than 50% papillary serous or clear cell histology on pathologic specimen
* Prior hysterectomy (total abdominal, vaginal hysterectomy, or laparoscopic-assisted vaginal hysterectomy) and bilateral salpingo-oophorectomy with or without additional surgical staging for endometrial cancer no more than 8 weeks prior to study
* No known metastatic extrauterine metastases, known gross residual disease, positive peritoneal cytology, or distant metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,800/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No cardiac dysrhythmias

Other:

* No other malignancy within the past 5 years except nonmelanomatous skin cancer
* No medical contraindications to study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M. Greven, MD, Study Chair — Wake Forest University Health Sciences; Richard R. Barakat, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (29):
- United States (28):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Brookview Research, Inc., Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Norwegian Radium Hospital, Oslo, Norway